CLINICAL TRIAL: NCT06605612
Title: Development and Validation of the FBIndex to Determine the Risk of Falls for Patients With Neuromuscular Disorders
Acronym: FBIndex
Status: Enrolling by invitation | Type: Observational
Sponsor: LMU Klinikum (Other)
Collaborators: Medical Park AG (Industry)
Responsible Party: Principal Investigator, Marko Mijic, Scientific Worker (dr. rer. biol. hum.), LMU Klinikum
Other Study IDs: 24-0636; 24-0636 (Other: Ludwig-Maximilians-Universität München / Ethikkommission)
Record Dates: First submitted 2024-09-09; First posted 2024-09-20 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Inclusion Body Myositis; Myotonic Dystrophy; Limb-girdle and Facioscapulohumeral Muscular Dystrophies; Pompe Disease; Myasthenia Gravis; Lambert-Eaton-Syndrome; Amyotrophic Lateral Sclerosis; Spinal Muscular Atrophy; Guillain-Barré Syndrome; Chronic Inflammatory Demyelinating Polyneuropathy; Friedreich Ataxia; Hereditary Motor Sensory Neuropathy
Keywords: Risk of falls; Neuromuscular Diseases; Neuromuscular Disorders; Risk of Falls Index; Assistive Gait Device
MeSH Terms: conditions — Myositis, Inclusion Body; Myotonic Dystrophy; Muscular Dystrophy, Facioscapulohumeral; Glycogen Storage Disease Type II; Myasthenia Gravis; Lambert-Eaton Myasthenic Syndrome; Amyotrophic Lateral Sclerosis; Muscular Atrophy, Spinal; Guillain-Barre Syndrome; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Friedreich Ataxia; Hereditary Sensory and Motor Neuropathy; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Friedrich-Baur-Institute: All patients in group A will undergo single tests (cross-over design data):HRT, CRT, STS, FTT and TRT on the Leonardo Mechanograph® Ground Reaction Force Plate, assessing power and force data. Additionally, the time to perform the tests will be assessed manually. The 10MWT, 6MWT and TUG tests are performed without a ground reaction force plate and only time parameters are assessed. The group A will have an additional subgroup A1 of n=20 patients, which will be tested two times within two weeks to confirm intra-rater (n=10) and inter-rater reliability (n=10).No intervention will be carried out.
  Interventions: Diagnostic Test: FBIndex
- Medical Park Bad Feilnbach: The group B will perform the same tests without using a force plate, assessing only the time parameters. No intervention will be carried out.
  Interventions: Diagnostic Test: FBIndex

INTERVENTIONS:
Diagnostic Test: FBIndex — There will be no intervention.

SUMMARY:
Currently, there are no standardised fall risk scores or guidelines on when to use appropriate assistive gait devices (AGDs) for people with neuromuscular disorders (NMDs). There is a clear medical unmet need to provide a battery of appropriate locomotor gait assessments to determine the risk of falling for patients with NMDs and give clear guidelines to prescribe an appropriate AGD.

The primary goal is to confirm whether the clinical battery assessments (Heel-Rise Test (HRT), Chair-Rise Test (CRT), Semi-tandem Stand (STS), Trunk-Rise Test (TRT), Foot-Tapping Test (FTT), Timed Up and Go (TUG), 10-Meter-Walk Test (10MWT) and 6-Minute-Walk Test (6MWT) can be validated and generalized to other NMD target populations that meet broader eligibility criteria based on used clinical assessments. The second objective of this project is to provide intra- and inter-observer reliability and test-retest reliability of included clinical assessments used to determine the risk of falling for patients with NMDs. Finally, all data will be compared with norm data from the healthy population (n=15) collected retrospectively.

DETAILED DESCRIPTION:
The NMD people are characterised by a complex muscle weakness caused by a combination of different factors. These include reduced endurance, lack of explosive muscle force and power, intramuscular strength coordination, and reduced balance. Those parameters need to be considered when developing an appropriate fall risk score. The combination of short muscular function and balance assessments with short clinical scores, can be a new, valid approach to evaluating the patient's risk of falling. In addition, it assists in creating a quick checkup for prescribing an appropriate assistive device.

In the first part (feasibility study) of this project, the following force plate tests were identified as suitable to assess muscle power, force and balance variables: Heel-Rise Test (HRT), Chair-Rise Test (CRT), Semi-tandem Stand (STS), Trunk-Rise Test (TRT), Foot-Tapping Test (FTT). They were used as predictors to assess patients muscle weakness and disability. In addition to muscle power and force data collected on the force plate, a second rater manually evaluated the time required to perform this test using a stopwatch. Additionally, three separate tests, Timed Up and Go (TUG), 10-Meter-Walk Test (10MWT) and 6-Minute-Walk Test (6MWT), have been evaluated separately as standard care procedures. The TUG, 10MWT and 6MWT have been used to assess remaining motor skills (endurance, walking speed and coordination) that cannot be covered by HRT, CRT, STS, TRT and FTT. As a third parameter used for correlation analysis, two risk of fall scales, Falls Efficacy Scale International (FES-I) and Morse Fall Scale (MFS), have been used. The found data from the feasibility study, which is planned to be published, suggest a moderate to moderate to strong correlation between HRT, CRT, STS, TRT, FTT, TUG, 10MWT and 6MWT and the FES-I and will be used in in the follow-up study. The MFS was excluded from the final test battery due to a lack of correlation with dependent variables. Moreover, the dependent variables assessed on the force plate, HRT, CRT, STS, TRT, and FTT (power and force), were correlated with variables collected by performing the same test using only manual time. Applying muscle strength and power data on the force plate was necessary to confirm internal consistency, content and criterion validity, as well as the degree to which the HRT, CRT, STS, TRT and FTT test can be an adequate reflection of the same test data using only manual time variables, as the final Friedrich-Baur Risk of Fall Index (FBIndex) should be conducted without the force plate using only time variables.

This study decided to include more patients and more different neuromuscular diseases to assess a wider range of muscle weaknesses that can lead to falls. Moreover, the final test battery was defined, and the standardised methodological procedure was established.

Using regression and discrimination analysis, the cross-sectional construct validity of a priori hypotheses: "Is there a multiple correlation between HRT, CRT, STS, TRT, FTT, TUG, 10MWT and 6MWT with FES-I?" will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Only patients with adequate cognitive and communicative function to give informed consent and to fill out the scale assessing the risk of falling will be included.

Exclusion Criteria:

* Patients who are unable to walk without AGD for at least 10 meters.
* Patients who had knee, hip or back surgery in the last three months.
* Patients who suffer from polyneuropathy or peripheral neuropathy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Following neuromuscular diseases confirmed by the genetic report and/or clinical final diagnosis will be included in the study: inclusion body myositis, myotonic dystrophies, limb-girdle and facioscapulohumeral muscular dystrophies, Pompe disease, myasthenia gravis, Lambert-Eaton-Syndrome, amyotrophic lateral sclerosis, spinal muscular atrophy, Guillain-Barré syndrome, chronic inflammatory demyelinating polyneuropathy, Friedreich-Ataxia, hereditary motor sensory neuropathy.
Sampling Method: Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Chair-Rise Test (CRT) | Immediately after the ICF is signed
  This is a sit-to-stand test with five repetitions. Three sets will be performed, and the fastest one will be scored. In Group A, the test uses a bench with a height of 46 cm anchored to the force plate.Only the best rise will be analyzed to collect force and power data. The main outcome parameter is the time required to perform the five repeat movements. In Group A, the examiner will assess the performance time of five sit-to-stand movements from the first to last repetition and the power data (Pmax rel. W/kg) from the force plate. In Group B, the examiner will only record the time taken to complete the test.
Trunk Rise Test (TRT) | Immediately after the ICF is signed
  Participants slowly bend their knees with erect straight upper body until the fingertips touch their feet or lower leg on the inside and then cross the arms on their chest and grab their shoulders with their hands. The instructions will follow: "After the signal, rise as fast as possible, one time (movement compared to lifting a heavy object). You can use your arm to push yourself up on your thigh if you cannot get up without it". Three sets will be done, and the fastest result will be evaluated. In Groups A and B, the examiner will assess the performance time from the start position "forward bend 90°" to stand up straight and also assess whether participants use their arms or not to stand up straight. In Group A, time is assessed with power data (Pmax rel. W/kg) from the force plate. In Group B, the examiner will only record the time to perform the test on a solid concrete ground floor.
Heel-Rise Test (HRT) | Immediately after the ICF is signed
  It consists of five bilateral maximal heel rises to achieve a maximal speed of upward movement. Three sets will be done, and the fastest result will be evaluated. The instructions will follow: "Rise to the tip of your toes five-times in a row as fast and high as possible. It is important that you keep your knees straight. Cross your arms on your chest and grab your shoulders with your hands. Move to your tiptoes as fast and high as possible." In Group A, the examiner will assess the performance time of five bilateral heel rises from first to last, along with the power data (P.max rel. kg- W/kg) from the force plate. In Group B, the examiner will only record the time to perform five bilateral heel rises from first to last tiptoes on a solid concrete ground floor.
Semi-Tandem stand, eyes open (STSeo) and eyes closed (STSeo) | Immediately after the ICF is signed
  In this test, participants will be instructed to stand as still as possible in an upright position with both arms crossed in front of the upper body for starting, first with eyes open. Then eyes closed, in a Semi-Tandem stand as long as possible (for a maximum of 30 sec.). Three sets will be done. During the test, the Leonardo Mechanography system records the position of the center of pressure on the platform. In Group A, the time to the first drop or side-step is measured, up to a maximum of 30 seconds, together with power data (Ellip. Average cm) from the force plate. In Group B, the examiner records only the time to first drop or side-step, up to a maximum of 30 seconds. The Group B will do a semi-tandem stand on a solid concrete floor with a 1 cm wide line between the inside of the soles of the feet.
Foot-Tapping Test (FTT) (sitting) | Immediately after the ICF is signed
  The FTT is designed to assess coordination and reaction time for the foot. Sitting on a 46 cm high bench, the participant's task is to tap ten times with the same foot (dorsal flexion, plantar flexion) as quickly as possible while keeping the heel on the ground. The participants were instructed to tap first with their right foot 10 times as quickly as possible. The same procedure will be repeated with the left feet, and three sets of left/right will be carried out. The participants need to sit straight, with 90° between the lower and upper leg and crossed arms over the chest. In Group A, the time for 10- foot tappings together with power data (max frequency and average contact time) from the force plate will be assessed. In Group B, the examiner records only the time. In Group B, participants are seated on a 46 cm high bench or chair with no backrest.
10-Meter Walk Test | Immediately after the ICF is signed
  Walking at maximum speed will be measured in a long corridor with an even surface over 10 meters with a still-standing start and a "flying" finish to a target 2.5 meters beyond the 10 m mark. The stopwatch started with the word "Go" ("Ready-Steady-Go").
Six-Minute Walk test | Immediately after the ICF is signed
  For the 6MWT, the individuals will be instructed to walk 30 m between two marks on the floor. After passing either mark, they will be told to turn and walk back. They will be instructed to walk as far as possible for six minutes and were allowed to rest (only while standing) and then to continue walking. They will be informed every minute of the remaining test time.
Time Up and Go (TUG) | Immediately after the ICF is signed
  The TUG test measures the time it takes to stand up from a chair, walk three meters, turn around and sit down in the same chair. The subjects start with arm support from a seated position in a chair of normal height (44-45 cm) with arms, walk at a comfortable and safe pace to a mark on the floor 3 meters away, turn around, walk back to the chair, turn again and sit down. Time is measured from the start of the moment until participants touch the chair backrest with their back.

SECONDARY OUTCOMES:
The Falls Efficacy Scale-International (FES-I) | Immediately after the ICF is signed
  FES_I, a valid and reliable risk of fall scale used for different diagnoses, will be performed. The patient will carry out the FES-I independently. The FES-I is a scale used to measure fear of falling, self-efficacy, and balance confidence. It is suitable for use in research and clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Friedrich-Baur-Institut, Neurologische Klinik und Poliklinik, LMU Klinikum, Ludwig-Maximilians-Universität München, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Undecided: It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Dias N, Kempen GI, Todd CJ, Beyer N, Freiberger E, Piot-Ziegler C, Yardley L, Hauer K. [The German version of the Falls Efficacy Scale-International Version (FES-I)]. Z Gerontol Geriatr. 2006 Aug;39(4):297-300. doi: 10.1007/s00391-006-0400-8. German. PMID 16900450
- [Background] Yardley L, Beyer N, Hauer K, Kempen G, Piot-Ziegler C, Todd C. Development and initial validation of the Falls Efficacy Scale-International (FES-I). Age Ageing. 2005 Nov;34(6):614-9. doi: 10.1093/ageing/afi196. PMID 16267188
- [Background] DiPaolo G, Jimenez-Moreno C, Nikolenko N, Atalaia A, Monckton DG, Guglieri M, Lochmuller H. Functional impairment in patients with myotonic dystrophy type 1 can be assessed by an ataxia rating scale (SARA). J Neurol. 2017 Apr;264(4):701-708. doi: 10.1007/s00415-017-8399-x. Epub 2017 Feb 6. PMID 28168524
- [Background] Murphy SM, Herrmann DN, McDermott MP, Scherer SS, Shy ME, Reilly MM, Pareyson D. Reliability of the CMT neuropathy score (second version) in Charcot-Marie-Tooth disease. J Peripher Nerv Syst. 2011 Sep;16(3):191-8. doi: 10.1111/j.1529-8027.2011.00350.x. PMID 22003934
- [Background] Runge M, Hunter G. Determinants of musculoskeletal frailty and the risk of falls in old age. J Musculoskelet Neuronal Interact. 2006 Apr-Jun;6(2):167-73. PMID 16849828
- [Background] Dharmadasa T, Matamala JM, Huynh W, Zoing MC, Kiernan MC. Motor neurone disease. Handb Clin Neurol. 2018;159:345-357. doi: 10.1016/B978-0-444-63916-5.00022-7. PMID 30482326